CLINICAL TRIAL: NCT01457222
Title: Mindfulness as a Method of Improving Mental Health and Cognitive Results and Decreasing Stress in Secondary School Students; a Prospective Randomised Controlled Single-blinded Pilot Study
Brief Title: Cognition and Health in Adolescents, Mindfulness as Prevention of Stress.
Acronym: CHAMPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2011/345
Record Dates: First submitted 2011-10-10; First posted 2011-10-21 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Stress; Complete Psychological Check Up; Sleep; Cognition - Other; Personality
Keywords: Mindfulness; Stress; Cognition; Psychological health; Primary prevention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness (Active Comparator): Mindfulness intervention 10 minutes daily
  Interventions: Behavioral: Mindfulness intervention
- Music relaxation (Active Comparator): Music intervention 10 minutes daily
  Interventions: Behavioral: Music relaxation
- Business as usual (No Intervention): No intervention - control group.

INTERVENTIONS:
Behavioral: Mindfulness intervention — Web-based guided mindfulness meditation 10 minutes daily
  Other Names: Mindfulnesscenter, Web-based mindfulness intervention
  Arms: Mindfulness
Behavioral: Music relaxation — Music relaxation 10 minutes daily
  Other Names: Music relaxation by Paxx
  Arms: Music relaxation

SUMMARY:
The purpose of this study is to determine whether mindfulness is useful as primary prevention for psychological health in highschool students, primarily related to stress, and whether mindfulness can improve cognitive function.

DETAILED DESCRIPTION:
There is a general suspicion that stress and stress-related psychological disorders is growing in highschool students in Sweden. Mindfulness is a well researched therapeutical method for treating stress-related disorders. This study will first collect data on stress-related psychological symptoms by several well-validated surveys. The surveys will be made twice with 8 weeks in between to examine variability. After the second survey the population of highschool students will be randomly assigned to web-based mindfulness intervention, music relaxation intervention or control group. A third survey will be conducted after eight weeks of intervention and before and after an external stressor.

ELIGIBILITY:
Inclusion Criteria:

* High school student from designated school

Exclusion Criteria:

* None Swedish-speaking

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Better mental health | Baseline to Eight weeks
  Lower Global Severity Index (from SCL-90) intrapersonal change

SECONDARY OUTCOMES:
Better sleep quality | Baseline to Eight weeks
  Lower result on Pittsburgh Sleep Quality Index
Lower degree of perceived stress | Baseline to Eight weeks
  Lower result on Perceived Stress Scale
Cognitive enhancement | Baseline to Eight weeks
  Shorter time on Trailmaking A and B as well as higher result on Symbol-Digit
Higher grades | Baseline to 6 months
  Higher mean school grades
Lower sick leave | Baseline to 6 months
  Less days of sick leave
Lower Neuroticism | Baseline to Eight weeks
  Lower Neuroticism result on Eysenck's Personality Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sundquist, Professor/MD, Study Chair — Centrum för Primärvårdsforskning
Locations (1):
- Centrum för Primärvårdsforskning, Lunds Universitet, Malmo, Sweden